CLINICAL TRIAL: NCT02405299
Title: Evaluation Des rééducations Neuropsychologiques Des Troubles de l'Inhibition Chez l'Enfant Avec un TDAH
Brief Title: Assessment of Neurocognitive Rehabilitations of Inhibition of Disorders in ADHD in Children (ERNTITDAH)
Acronym: ERNTITDAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L'hôpital Nord-Ouest - Villefranche Villefranche sur Saône (Other)
Responsible Party: Principal Investigator, Coline Perrier, Ms. Seguin Charlotte, neuropsychologist psychologist, L'hôpital Nord-Ouest - Villefranche Villefranche sur Saône
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HNOVillefranche
Record Dates: First submitted 2014-12-12; First posted 2015-04-01 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: ADHD
Keywords: child; disorders inhibition; neuropsychology; rehabilitation; ADHD; assessment of neurocognitive rehabilitations in ADHD in children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): neuropsychological reeducation disorder specific of inhibition (bottom-up and top-down protocol): 24 bi-weekly sessions (30 subjects)
  Interventions: Other: experimental groupe
- Control Group (Placebo Comparator): non-specific and general cognitive neuropsychological reeducation (comprehension, syntactic, visuospatial) : 24 bi-weekly sessions (30 subjects)
  Interventions: Other: experimental groupe

INTERVENTIONS:
Other: experimental groupe — exercices of cognitive and neuropsychological stimulation of inhibition (paper and pencil exercises and computerized exercises) created for the experience: cognitive stimulation exercises for children in the form of cognitive and metacognitive games with rehabilitation objective disorder of inhibition

SUMMARY:
This research aims to assess the cognitives rehabilitations in attention deficit disorder (ADHD) in children. the objective is to demonstrate what are the most relevant cognitive factors for rehabilitative to improve the inhibition of disorders in ADHD.

DETAILED DESCRIPTION:
This study examines the effect of neuropsychological rehabilitation on the disorder inhibtion in the child with ADHD.

Sample includes 60 subjects aged 9-13 years with disorder of inhibition evalued with neuropsychological test. Neuropsychological rehabilitation protocol was developed and evaluated.

This study use baseline and includes a control group and an experimental group. The type of cognitive procedure (up / down, or rehabilitative / metacognitive) is examined.

ELIGIBILITY:
Inclusion Criteria:

* presence of a disorder of inhibition (assessed by neuropsychological subtests) as part of an ADHD with normal intellectual potential (ICV WISC4) in children born at term or preterm (-33SA)

Exclusion Criteria:

* patient refusal and family to participate in the study
* subjects with sensory disorders, psychological or unsupported, subjects carrying other cognitive disorders prevalent disorder of inhibition
* subjects with psychostimulant treatment at inclusion in the study

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
scores to neuropsychological testing inhibition before and after rehabilitation in experimental groupe | 5 months
  comparison of the results obtained by the experimental subjects neuropsychological tests before and after rehabilitation (standard notes to NEPSY subtests, TAP, TEA-ch, Stroop test)

SECONDARY OUTCOMES:
scores to neuropsychological testing inhibition before and after rehabilitation in control group | 5 months
  comparison of the results obtained by the control group subjects neuropsychological tests before and after rehabilitation (standard notes to NEPSY subtests, TAP, TEA-ch, Stroop test)

CONTACTS AND LOCATIONS:
Locations (1):
- Seguin, Villefranche-sur-Saône, Rhone, France